CLINICAL TRIAL: NCT02391090
Title: Effects of Intermittent Hypoxia on the Asthmatic Inflammation of Asthma Patients - a Pilot Study
Brief Title: FeNO After Hypoxia in Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Ludwig Boltzmann Institute for Lung Vascular Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MUG-FeNO-2013
Record Dates: First submitted 2015-01-26; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Asthma
Keywords: asthma; hypoxia; forced exhaled nitric oxide; inflammation
MeSH Terms: conditions — Asthma; Hypoxia; Inflammation | interventions — Oximetry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypoxia (Experimental): The hypoxia group receives normobaric hypoxic air while sitting in a hypoxic chamber simulating 2800 meter above sea level.
  Interventions: hypoxia in hypoxic chamber, asthma and Quality of Life Questionnaires, lung function testing, blood taking, FeNO measurement, pulse oximetry
  Interventions: Device: hypoxia in hypoxic chamber; Procedure: Pulse oximetry; Other: Asthma and Quality of Life Questionnaires; Procedure: Lung function testing; Procedure: Blood taking; Procedure: FeNO measurement
- sham hypoxia (Sham Comparator): The sham group receives normal air while sitting in a hypoxic chamber in about 360 meter above sea level (Graz, Austria).
  Interventions: sham hypoxia in hypoxic chamber, asthma and Quality of Life Questionnaires, lung function testing, blood taking, FeNO measurement, pulse oximetry
  Interventions: Device: sham hypoxia in hypoxic chamber; Procedure: Pulse oximetry; Other: Asthma and Quality of Life Questionnaires; Procedure: Lung function testing; Procedure: Blood taking; Procedure: FeNO measurement

INTERVENTIONS:
Device: hypoxia in hypoxic chamber — Intervention lasts 4 hours per day for 6 days in a row.
  Arms: hypoxia
Device: sham hypoxia in hypoxic chamber — Intervention lasts 4 hours per day for 6 days in a row.
  Arms: sham hypoxia
Procedure: Pulse oximetry — Pulse oximetry will be performed hourly during sessions in the hypoxic chamber for safety reasons.
Other: Asthma and Quality of Life Questionnaires — Before every session in the hypoxic chamber as well as on the day after the last session will be completed.
Procedure: Lung function testing — On the day of the first session in the hypoxic chamber as well as on the day after the last session lung function testing will be performed.
Procedure: Blood taking — On the day of the first session in the hypoxic chamber as well as on the day after the last session blood samples will be taken.
Procedure: FeNO measurement — Before every session in the hypoxic chamber as well as on the day after the last session FeNO (forced exhaled nitric oxide) measurement will be performed.

SUMMARY:
Stable Asthma patients (GINA 1-2) stay 6 days in a row for 4 hours per day in a hypoxic chamber simulating 2800m above sea level. Study participants will be blinded to the treatment given and divided into a hypoxic and a sham group (about 360m above sea level).

Effects of this intermittent hypoxia on the asthmatic inflammation of these patients will be measured. The primary endpoint is the change in forced exhaled nitric oxide (FeNO) before and after the study. Secondary endpoints include blood parameters, lung function testing and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* stable Asthma (GINA 1-2)

Exclusion Criteria:

* autoimmune disease
* unstable Asthma (GINA 3-4)
* history of pneumonia/fever within 3 months
* place of residence >1000m above sea level
* trip/vacation above >2500m within 4 weeks
* cystic fibrosis
* diabetes mellitus
* immunodeficiency
* atopic dermatitis
* ciliary dyskinesia
* pregnancy
* chronic obstructive pulmonary disease
* history of smoking (>1py)
* immunosuppression / systemic corticosteroids within 3 months
* cardiovascular diseases
* interstitial lung disease
* bronchopulmonary dysplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in forced exhaled nitric oxide after 6 days of hypoxia/sham | 1 week
  Forced exhaled nitric oxide will be measured every day before and after the treatment

SECONDARY OUTCOMES:
Change in blood parameters after 6 days of hypoxia/sham | 1 week
  Blood parameters including c-reactive protein, complete blood cell count, total immunoglobulin e (IgE), specific IgE of seasonal inhalative antigens and eosinophilic cationic protein will be measured. Blood samples will be taken before the first and after the last intervention
Change in lung function parameters after 6 days of hypoxia/sham | 1 week
  Lung function testing will be performed before the first and after the last intervention
Change in Quality of Life and Asthma questionnaires after 6 days of hypoxia/sham | 1 week
  Questionnaires include Asthma Control Test, Asthma Quality of Life Questionnaire, Asthma Control Questionnaire, a quality of life questionnaire and the Asthma Control Diary. Documents will be collected every day before the intervention
Change in finger pulse oximetry | 1 week
  Finger pulse oximetry will be measured hourly during the intervention for safety reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Prof., Principal Investigator — Medical University of Graz, Department of Internal Medicine, Division of Pulmonology
Locations (1):
- Medical University of Graz, Graz, Styria, Austria